CLINICAL TRIAL: NCT05358730
Title: Instrument-assisted Soft Tissue Mobilization to Exercise Programme Improves Outcomes in Patients with Adhesive Capsulitis
Brief Title: Effects of IASTM in the Treatment of Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, Tansu Birinci, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1008
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2022-05

CONDITIONS: Pain, Shoulder; Adhesion; Shoulder; Myofacial Pain
Keywords: Adhesive capsulitis; Function; Pain; Exercise
MeSH Terms: conditions — Shoulder Pain; Tissue Adhesions; Facial Pain; Bursitis; Pain; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IASTM + Standard Exercise Group (Experimental): Patients were applied IASTM in combination with standard exercise program two days a week for six weeks. The IASTM technique was performed using six titanium-plated instruments in different sizes, shapes and treatment styles. ROM, crutch, roller, scapulothoracic and stretching exercises were given as home exercises during the treatment.
  Interventions: Other: Standard Exercise; Other: Instrument Assisted Soft Tissue Mobilization (IASTM); Other: Home Exercise
- Standard Exercise Group (Active Comparator): Patients were given a standard exercise program two days a week for six weeks. ROM, crutch, roller, scapulothoracic and stretching exercises were given as home exercises during the treatment.
  Interventions: Other: Standard Exercise; Other: Home Exercise

INTERVENTIONS:
Other: Standard Exercise — Glenohumeral exercises, scapulothoracic exercises, stretching exercises and mobilization exercises were performed under the supervision of a physiotherapist two days per week for six weeks at the clinical setting (Celik and Kaya Mutlu, 2016).
Other: Instrument Assisted Soft Tissue Mobilization (IASTM) — IASTM treatment was applied to the posterior-anterior-middle deltoid, latissimus dorsi, teres major, teres minor, supraspinatus and infraspinatus muscle fibers, superficial and deep fascia. IASTM was applied in parallel and vertical direction to the muscle fibers treated with the instrument at a 45° angle, each technique (SWEEP, BRUSH (straight short steps) techniques) for 20 seconds (Ikeda, Otsuka, Kawanishi, and Kawakami, 2019). It was performed two days per week for six weeks.
  Arms: IASTM + Standard Exercise Group
Other: Home Exercise — Hme exercise program consisted of glenohumeral exercises, scapulothoracic exercises, stretching exercises and mobilization exercises.
  It was asked to perform two days per week for six weeks.

SUMMARY:
This study aimed to determine the effects of IASTM in combination with exercise in frozen shoulder. Thirty-five patients with phase II frozen shoulder included in this single-blind, randomized study. Patients were divided into two groups. In the first group exercise programme (Group 1) and in the second group IASTM in combination with exercise programme (Group 2) were applied for twelve sessions (two days per week for six week). The primary outcome was the Disabilities of the Arm, Shoulder and Hand (DASH) score and secondary outcomes were the visual analogue scale (VAS), the range of motion (ROM), The Constant score and Short- Form-36 (SF-36). Outcome measures were performed at baseline, after the 6th session and the 12th session.

DETAILED DESCRIPTION:
Instrument Assisted Soft Tissue Mobilization (IASTM) is a popular treatment for myofascial restriction based on the logic developed by James Cyriax. IASTM is applied using specially designed instruments to provide a mobilizing effect on soft tissue (eg scar tissue, myofascial adhesion) to reduce pain, improve joint range of motion and function. IASTM can help improve fibroblast proliferation and promote normal collagen sequencing, however, there is no enough study evaluating the results of IASTM use in patients with frozen shoulders in the literature. This study aimed to determine the effects of IASTM in combination with exercise in the treatment of frozen shoulder. Therefore, it was hypothesized that exercise programme combined with IASTM are more effective in improving pain, range of motion (ROM), and functionality than are the exercise programme alone.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 30 and 65 years;
* Duration of complaint of more than three months
* ROM in external rotation, abduction and flexion less than 50% in comparison to uninvolved shoulder in one or more of three movement directions

Exclusion Criteria:

* Having cervical radiculopathy
* Thoracic outlet syndrome
* Rheumatological disorders
* Fractures or tumors of either upper extremity
* Corticosteroid injections in the affected shoulder within the previous 4 weeks

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2019-08-10 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Upper extremity function | Baseline
  DASH is a 30-item questionnaire that evaluates functionality, pain, emotional and social parameters in the upper extremity. Twenty-one questions evaluate patients' difficulties in daily life activities, 5 questions symptoms, 4 questions social function, work, sleep and self-confidence. For each question, the participant marks the option that suits patients in the 5-point Likert system (1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: inability). Score between 0 and 100 were obtained from each section.

SECONDARY OUTCOMES:
Upper extremity function | At the end of the 3-week intervention
  DASH is a 30-item questionnaire that evaluates functionality, pain, emotional and social parameters in the upper extremity. Twenty-one questions evaluate patients' difficulties in daily life activities, 5 questions symptoms, 4 questions social function, work, sleep and self-confidence. For each question, the participant marks the option that suits patients in the 5-point Likert system (1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: inability). Score between 0 and 100 were obtained from each section.
Upper extremity function | At the end of the 6-week intervention
  DASH is a 30-item questionnaire that evaluates functionality, pain, emotional and social parameters in the upper extremity. Twenty-one questions evaluate patients' difficulties in daily life activities, 5 questions symptoms, 4 questions social function, work, sleep and self-confidence. For each question, the participant marks the option that suits patients in the 5-point Likert system (1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: inability). Score between 0 and 100 were obtained from each section.
The severity of pain | Baseline
  The severity of pain that people feel on their shoulders at rest, during activity and at night was evaluated using the Visual Analogue Scale (VAS). The patients were told that "0" number shows "no pain" and "10" number shows "most excruciating pain" on the visual analog scale, and the participant was asked to position the pain feeling in this range by drawing a line.
The severity of pain | At the end of the 3-week intervention
  The severity of pain that people feel on their shoulders at rest, during activity and at night was evaluated using the Visual Analogue Scale (VAS). The patients were told that "0" number shows "no pain" and "10" number shows "most excruciating pain" on the visual analog scale, and the participant was asked to position the pain feeling in this range by drawing a line.
The severity of pain | At the end of the 6-week intervention
  The severity of pain that people feel on their shoulders at rest, during activity and at night was evaluated using the Visual Analogue Scale (VAS). The patients were told that "0" number shows "no pain" and "10" number shows "most excruciating pain" on the visual analog scale, and the participant was asked to position the pain feeling in this range by drawing a line.
Functional level of shoulder | Baseline
  The modified constant shoulder score assesses pain, position, daily living activities, ROM and strength. Scoring consists of pain (15 points), daily activities (20 points), active range of motion (AROM) (40 points) and strength (25 points). The total Constant score is classified as excellent (90-100), good (80-89), moderate (70-79) and poor (<70). Turkish validity and reliability study of modified constant score.
Functional level of shoulder | At the end of the 3-week intervention
  The modified constant shoulder score assesses pain, position, daily living activities, ROM and strength. Scoring consists of pain (15 points), daily activities (20 points), active range of motion (AROM) (40 points) and strength (25 points). The total Constant score is classified as excellent (90-100), good (80-89), moderate (70-79) and poor (<70). Turkish validity and reliability study of modified constant score.
Functional level of shoulder | At the end of the 6-week intervention
  The modified constant shoulder score assesses pain, position, daily living activities, ROM and strength. Scoring consists of pain (15 points), daily activities (20 points), active range of motion (AROM) (40 points) and strength (25 points). The total Constant score is classified as excellent (90-100), good (80-89), moderate (70-79) and poor (<70). Turkish validity and reliability study of modified constant score.
Range of motion | Baseline
  Shoulder flexion, abduction, internal rotation and external rotation ROM were actively and passively measured using a universal goniometer while the participant was in the supine position. All shoulder ROMs were repeated 3 times and the average of the angular values obtained was recorded in degrees.
Range of motion | At the end of the 3-week intervention
  Shoulder flexion, abduction, internal rotation and external rotation ROM were actively and passively measured using a universal goniometer while the participant was in the supine position. All shoulder ROMs were repeated 3 times and the average of the angular values obtained was recorded in degrees.
Range of motion | At the end of the 6-week intervention
  Shoulder flexion, abduction, internal rotation and external rotation ROM were actively and passively measured using a universal goniometer while the participant was in the supine position. All shoulder ROMs were repeated 3 times and the average of the angular values obtained was recorded in degrees.
Health-related quality of life | Baseline
  In order to evaluate the quality of life, the Short Form-36 (SF-36) was used, which consists of 36 items evaluating 2 main (physical and mental component) and 8 sub-parameters (physical, emotional and social function, physical role, mental health, pain, general health and vitality). The scale evaluating the score of each subgroup between 0-100; 0 indicates "bad health", 100 indicates "good health". In our study, SF-36 health control scale scoring was calculated on the internet address http://www.rand36calculator.com with the percentage values given as a result of marking the answers in the form.
Health-related quality of life | At the end of the 3-week intervention
  In order to evaluate the quality of life, the Short Form-36 (SF-36) was used, which consists of 36 items evaluating 2 main (physical and mental component) and 8 sub-parameters (physical, emotional and social function, physical role, mental health, pain, general health and vitality). The scale evaluating the score of each subgroup between 0-100; 0 indicates "bad health", 100 indicates "good health". In our study, SF-36 health control scale scoring was calculated on the internet address http://www.rand36calculator.com with the percentage values given as a result of marking the answers in the form.
Health-related quality of life | At the end of the 6-week intervention
  In order to evaluate the quality of life, the Short Form-36 (SF-36) was used, which consists of 36 items evaluating 2 main (physical and mental component) and 8 sub-parameters (physical, emotional and social function, physical role, mental health, pain, general health and vitality). The scale evaluating the score of each subgroup between 0-100; 0 indicates "bad health", 100 indicates "good health". In our study, SF-36 health control scale scoring was calculated on the internet address http://www.rand36calculator.com with the percentage values given as a result of marking the answers in the form.

CONTACTS AND LOCATIONS:
Overall Officials: Tansu Birinci, PT, PhD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Bakırkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No